CLINICAL TRIAL: NCT02356692
Title: Clinical Comfort Evaluation of Two Marketed Spherical Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-38-MTF
Record Dates: First submitted 2012-04-30; First posted 2015-02-05 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- enfilcon A (Experimental): participants randomized to wear the Enfilcon A (test) lens in one eye and Senofilcon A (control) lens in the other eye.
  Interventions: Device: enfilcon A; Device: senofilcon A
- senofilcon A (Active Comparator): participants randomized to wear the Enfilcon A (test) lens in one eye and Senofilcon A (control) lens in the other eye.
  Interventions: Device: enfilcon A; Device: senofilcon A

INTERVENTIONS:
Device: enfilcon A — Test lens
Device: senofilcon A — Control lens

SUMMARY:
The purpose of this study was to investigate the overall clinical comfort performance of enfilcon A (test) lens and senofilcon A (control) lens over 15-minutes of lens wear.

DETAILED DESCRIPTION:
This was a non-dispensing, single-masked, randomized, contralateral study comparing Enfilcon A (test) against Senofilcon A (control). Each subject was randomized to wear the test lens in one eye and the control lens in the other eye.

ELIGIBILITY:
Inclusion Criteria:

1. Based on his/her knowledge, must be in good general health.
2. Be 18 to 38 years old.
3. Be able and willing to adhere to the instructions set forth in this protocol and complete all specified evaluation.
4. Read, indicate understanding of, and sign Written Informed Consent.
5. Be existing or successfully adapted users of soft contact lenses, but not currently wearing either of the study lenses (Avaira or Oasys) being evaluated in this trial.
6. Require a visual correction in both eyes.
7. Require a prescription between +8.00D and -12.00D and have less than or equal to 0.75D of astigmatism in both eyes.
8. Achieve visual acuity of 20/25 or better in each eye with a spherical contact lens prescription.
9. Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

   * No amblyopia.
   * No evidence of lid abnormality or infection (e.g. entropion, ectropion, chalazia, recurrent styes).
   * lamp findings Grade 2 or above: corneal edema, tarsal abnormalities, and conjunctival injection).
   * No other active ocular disease (e.g. glaucoma, history of recurrent corneal erosions, cornea [infiltrates], conjunctiva, lids, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology).
   * No aphakia.

Exclusion Criteria:

1. 0.75D or greater of refractive astigmatism in either eye.
2. Presbyopic or current monovision contact lens wear.
3. Cannot be currently wearing either lenses (Avaira or Oasys).
4. Presence of clinically significant (grade 2-4) anterior segment abnormalities; inflammation such as iritis; or any infection of the eye, lids, or associated structures.
5. Presence of ocular or systemic disease or need of medication which might interfere with contact lens wear.
6. Slit lamp findings that would contraindicate contact lens wear such as:

   * Pathological dry eye or associated findings
   * Pterygium, pinguecula or corneal scars within the visual axis
   * Neovascularization > 0.75 mm in from the limbus
   * Giant papillary conjunctivitis (GPC) worse than Grade 1
   * Anterior uveitis or iritis (past or present)
   * Seborrheic eczema, seborrheic conjunctivitis
   * History of corneal ulcer or fungal infections
   * Poor personal hygiene
   * A known history of corneal hypoesthesia (reduced corneal sensitivity)
7. Contact Lens best corrected Snellen visual acuities (VA) worse than 20/30.
8. Aphakia, Keratoconus or a highly irregular cornea.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Siegel, OD, Study Chair — CooperVision, Inc.
Locations (3):
- United States (3):
  - Schaeffer Eye Associates, Birmingham, Alabama
  - Beaches Family Eyecare, Jacksonville, Florida
  - Todays Eyecare, LLC, Lafayette, Louisiana

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Enfilcon A: participants randomized to wear the (enfilcon A) test lens in one eye.
  Enfilcon A: contact lens
- Senofilcon A: participants randomized to wear the senofilcon A contact lens (control) in the one eye.
  Senofilcon A: contact lens
Period: Overall Study
Arm/Group | Enfilcon A | Senofilcon A
Started | 60; 60 Eyes | 60; 60 Eyes
Completed | 60; 60 Eyes | 60; 60 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Group: participants randomized to wear the (enfilcon A) test lens in one eye and the senofilcon A (control) in the other eye.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Comfort at Insertion
Description: Participant's response for comfort at insertion. (Scale 0-10; 0=poor/intolerable, 10=comfortable/ cannot be felt) Obtained at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Senofilcon A: participants randomized to wear the senofilcon A (control) lens in the one eye.
  senofilcon A: contact lens
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 60 | 60
Number analyzed (eyes) | 60 | 60
units on a scale | 8.7 (1.6) | 8.5 (1.7)

2. Primary Outcome: Comfort at Insertion
Description: Participant's response for comfort at 15 minutes. (Scale 0-10; 0=poor/intolerable, 10=comfortable/ cannot be felt) Obtained at 15 minutes.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Senofilcon A: participants randomized to wear the senofilcon A control lens in one eye.
  senofilcon A: contact lens
Arm/Group | Enfilcon A | Senofilcon A
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
units on a scale | 8.1 (1.8) | 8.7 (1.3)

3. Primary Outcome: Comfort Preference
Description: Participant's response for comfort preference of enfilcon A (test) lens, senofilcon A(control) lens at insertion.
Time Frame: Baseline
Population: n=59, one participant would not choose a preference at the initial insertion as both lenses were the same to them.
Measure: Number; unit: participants
Groups:
- Overall Study Group: participants randomized to wear the (enfilcon A) test lens in one eye and the senofilcon A (control) in the other eye.
  Enfilcon A: contact lens Senofilcon A: contact lens
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
participants
  Prefer Enfilcon A | 30
  Prefer Senofilcon A | 29

4. Primary Outcome: Comfort Preference
Description: Participant's response for comfort of enfilcon A (test) lens, senofilcon A (control) lens at 15 minutes wear.
Time Frame: 15 minutes
Measure: Number; unit: participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
participants
  Preferred Enfilcon A | 25
  Preferred Senofilcon A | 35

ADVERSE EVENTS:
Time Frame: From dispense up to 15 minutes for both study lenses.
Groups:
- Enfilcon A: participants randomized to wear the test lens (enfilcon A) in one eye.
  Enfilcon A: contact lens
- Senofilcon A: participants randomized to wear the control lens (senofilcon A) in the one eye.
  Senofilcon A: contact lens
Arm/Group | Enfilcon A | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Recipient agress to maintain Confidential Information in strict confidence, not to disclose Confidential Information to any third parties and no to use Confidential Information for any purposes execpt for Business Purpose.